CLINICAL TRIAL: NCT03868852
Title: Efficacy and Safety of Radiotherapy Combined With Apatinib Mesylate in the Treatment of Rhabdomyosarcoma in Children
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XH-18-018
Record Dates: First submitted 2019-02-11; First posted 2019-03-11 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2019-02

CONDITIONS: Childhood Rhabdomyosarcoma
Keywords: Radiation Therapy; Rhabdomyosarcoma in Children
MeSH Terms: interventions — apatinib

STUDY DESIGN:
Intervention Model Description: Simons two-stage design method requires the enrollment of 13 patients in the first stage. If more than 7 patients fail to reach the expected end point, the first stage fails and the patients do not need to enter the second stage. A total of 48 patients were enrolled. If more than 30 patients did not reach the expected end point, the overall trial failed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiotherapy plus apatinib mesylate (Experimental): All eligible patients signed informed consent. Three-dimensional conformal intensity modulation (IMRT) technique was used to treat the patients with radiation doses 45 Gy - 54 Gy. All patients took apatinib mesylate tablets 250 mg QD orally from 1 week before radiotherapy to the whole radiotherapy period. They were required to take apatinib mesylate tablets with warm boiling water half an hour after meal. The daily medication time should be as consistent as possible.
  Interventions: Drug: Apatinib mesylate tablets; Radiation: Three-dimensional conformal intensity modulation

INTERVENTIONS:
Drug: Apatinib mesylate tablets — Apatinib mesylate tablets were orally administered 250 mg QD from 1 week before radiotherapy to the whole radiotherapy period. (Appatinib is no longer used after radiotherapy)
Radiation: Three-dimensional conformal intensity modulation — Three-dimensional conformal intensity modulation (IMRT) technique was used for post-operative radiotherapy. The radiation dose was 45-54 Gy.
  Other Names: 3D-IMRT

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of radiotherapy combined with apatinib mesylate in the treatment of rhabdomyosarcoma in children.

DETAILED DESCRIPTION:
This study is a Interventional study. The target group was 3-18 years old, and the pathological stage was group II-IV recurrence or distant metastasis. A total of 48 patients were enrolled in this study. The treatment was radiotherapy combined with apatinib. The main outcome measures were ORR, DCR , OS , quality of life and drug safety. The main safety indicators were vital signs, laboratory indicators, adverse events (AE), and severe adverse events (SAE). This study is expected to be enrolled for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥ 3 and ≤ 18 years of age.
* The predicted survival period is more than 3 months.
* According to RECIST version 1.1, there is at least one measurable lesion.
* Postoperative pathological stage was group II-IV.
* Patients have not received radiotherapy before, and can accept chemotherapy and surgical treatment.
* No other anticancer therapy should be used during radiotherapy.
* The main organs are functioning normally, which meets the following criteria:

  1. Blood routine examination standards should be met: (no blood transfusion within 14 days) A.HB>90g/L; B.ANC>1.5*109/L; C.PLT>80*109/L
  2. Biochemical tests should meet the following criteria:

A. BIL < 1.25 times normal upper limit (ULN); B. ALT and AST < 2.5 ULN; C. Serum Cr < 1 ULN, endogenous creatinine clearance > 50 ml/min

* Subjects volunteered to participate in this study, patients or legal guardians signed informed consent through patient consent, good compliance, with follow-up.
* Doctors believe that treatment can benefit patients.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | First analysis will occur 1 month after accrual of all patients.
  Refers to the proportion of patients whose tumors have shrunk to a certain extent and maintained for a certain period of time, including CR and PR cases. Objective remission of solid tumors was assessed by RECIST 1.1. Subjects must be accompanied by measurable tumor lesions at baseline. According to RECIST 1.1, the criteria for evaluating efficacy are complete remission (CR), partial remission (PR), stability (SD), and progression (PD).

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | First analysis will occur 1 month after accrual of all patients.
  The percentage of patients whose tumors shrink or remain stable for a certain period of time
Total Survival (OS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months.
  The time from enrollment to death for any reason. For those who had lost interviews before death, the last follow-up time was usually calculated as the time of death.
Quality of Life Score | Weekly assessment , assessed up to 1 month.
  Quality of life score refer to EORTC qlq-c30 (version 3, Chinese version). Quality of Life Questionnare-Core 30 prepared by The European O-rganization for Reasearch and Treatment of Cancer.
  EORTC qlq-c30 (V3.0) is the core scale for all cancer patients, with a total of 30 items. Items 29 and 30 are rated on a scale of 1 to 7 according to their answer choices. The other items are divided into four levels: totally not, a little bit, a lot and very much, and are scored on a scale of 1 to 4.
  The higher the score of functional domain and general health domain, the better the functional status and quality of life. The higher the score of symptom domain, the more symptoms or problems (the worse the quality of life).
Incidence and severity of Adverse Events | From date of enrollment until 30 days after the last medication.
  The safety of the drug was evaluated by NCI-CTCAE 4.0. Common Terminology Criteria Adverse Events Version 4.0 prepared by National Cancer Institute.

CONTACTS AND LOCATIONS:
Overall Officials: Mawei Jiang, MD, Principal Investigator — Xin Hua Hospital affiliated to Shanghai Jiaotong University School of Medicine
Locations (1):
- The Department of Radiation Oncology, Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vatner R, James CD, Sathiaseelan V, Bondra KM, Kalapurakal JA, Houghton PJ. Radiation therapy and molecular-targeted agents in preclinical testing for immunotherapy, brain tumors, and sarcomas: Opportunities and challenges. Pediatr Blood Cancer. 2021 May;68 Suppl 2:e28439. doi: 10.1002/pbc.28439. Epub 2020 Aug 22. PMID 32827353